CLINICAL TRIAL: NCT01775020
Title: Arginine and Nitric Oxide (NO) Metabolism in Sepsis; Dose-response Study on the Effect of L-arginine Supplementation on NO Metabolism and Gastric Perfusion in Severe Septic Patients.
Brief Title: Dose-response Study of Arginine Supplementation in Severe Sepsis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Novartis Medical Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MEC03-139.5
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-arginine (Experimental): L-arginine
  Interventions: Dietary Supplement: L-arginine

INTERVENTIONS:
Dietary Supplement: L-arginine
  Other Names: L-arginine-HCl

SUMMARY:
Pilot data in patients and data from pig studies indicate that arginine-NO metabolism is impaired in sepsis with changes in splanchnic metabolism and function, and reduced survival at low nitrate levels. Prolonged intravenous supplementation of L-arginine proved effective in pigs for increasing NO production, restoring gut function, and inhibiting an increase in pulmonary arterial pressure, without any deleterious systemic side effects. Prolonged intravenous L-arginine supplementation could therefore be useful in septic ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from close relative
* Age > 18 years
* Patient meets the general criteria for severe sepsis or septic shock, diagnosed less than 48 h prior to study inclusion (see appendix A; in Dutch).
* Patient must be relatively hemodynamically stable, defined as stable blood pressure (variation in mean arterial pressure <15 mm Hg) during 2 h without necessity of increasing the vasopressor dose, inotropic support or rate of fluid administration.
* Systemic and pulmonary arterial catheters in place with continuous pressure monitoring.
* Patients in whom the clinician is prepared to provide full life support during the duration of the study, including a life expectance of > 24 h.

Exclusion Criteria:

* Shock due to any cause other than sepsis (e.g. drug reaction or drug overdose, pulmonary embolus, burn injury etc.)
* Corticosteroid use (prolonged intake of > 1mg/kg daily or intake of > 70 mg/day for 7 consecutive days within 1 month preceding the study)
* Liver cirrhosis
* Chronic pancreatitis
* Diabetes mellitus type I
* Metastases, haematological malignancies or chemotherapy
* Patients on dialysis (CVVH or other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-10; Primary Completion 2004-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Nitric oxide synthesis | 8 hours
  Nitric oxide synthesis at step-wise increasing doses of L-arginine infusion. Following a 2h baseline measurements, 3 stepwise increasing arginine doses each provided for 2h will be tested for the effect on NO synthesis.

SECONDARY OUTCOMES:
hemodynamics | 8 hours
  Mean arterial pressure (MAP), pulmonary arterial pressure (PAP), cardiac output (CO), cardiac index (CI), heart rate (HR)
blood parameters | 8 hours
  Blood gasses, electrolytes, glucose, insulin, amino acids, whole body protein and arginine metabolism
gastric perfusion | 8 hours
  Regional (gastric) CO2 production measured with tonometry (PrCO2)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas E Deutz, MD PhD, Principal Investigator

REFERENCES:
- [Background] Luiking YC, Poeze M, Ramsay G, Deutz NE. Reduced citrulline production in sepsis is related to diminished de novo arginine and nitric oxide production. Am J Clin Nutr. 2009 Jan;89(1):142-52. doi: 10.3945/ajcn.2007.25765. Epub 2008 Dec 3. PMID 19056593
- [Background] Poeze M, Bruins MJ, Kessels F, Luiking YC, Lamers WH, Deutz NE. Effects of L-arginine pretreatment on nitric oxide metabolism and hepatosplanchnic perfusion during porcine endotoxemia. Am J Clin Nutr. 2011 Jun;93(6):1237-47. doi: 10.3945/ajcn.110.007237. Epub 2011 Apr 20. PMID 21508091